CLINICAL TRIAL: NCT05373459
Title: Effect of a Third COVID-19 Booster on COVID-19 Infection Rate and Return to Works During Fifth Wave COVID-19 Among Health Care Workers
Brief Title: Effect of a Third COVID-19 Booster Among Health Care Workers
Status: Completed | Type: Observational
Sponsor: Hong Kong Sanatorium & Hospital (Industry)
Responsible Party: Principal Investigator, Dr. Jonpaul ST Zee, Specialist in Infectious Disease, Hong Kong Sanatorium & Hospital
Other Study IDs: Third COVID-19 booster
Record Dates: First submitted 2022-05-12; First posted 2022-05-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: COVID-19 Vaccines
MeSH Terms: interventions — COVID-19 vaccine booster shot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health care workers without third COVID-19 booster: Health care workers received less than 3 doses of COVID-19 vaccine
- HCWs with third COVID-19 booster: Health care workers received at least 3 doses of COVID-19 vaccine
  Interventions: Biological: Third COVID-19 booster

INTERVENTIONS:
Biological: Third COVID-19 booster — Third COVID-19 booster
  Groups: HCWs with third COVID-19 booster

SUMMARY:
A new wave of COVID-19 infections, mainly caused by the Omicron/ Delta variant, has been sweeping the globe since the start of 2022. In response, the administration of a third dose of COVID-19 vaccine was considered to address potential waning immunity over time and reduced effectiveness against the Omicron/ Delta variant. The pandemic also resulted in many infections among health care workers (HCWs) and their households. In this study, a retrospective analysis would perform on risk of COVID-19 infection and their outcome in relation to their COVID-19 vaccination history by using the data repository from one of the Hong Kong private hospitals.

HCWs were required to submit a standardized online self-declaration form for report of 1) demographic of the HCWs, 2) symptoms related history and 3) COVID-19 exposure history once they were COVID-19 confirmed by rapid antigen test against COVID-19 and/or polymerase chain reaction (PCR) test for COVID-19. Subsequent follow up such as contact tracing, COVID-19 PCR testing results of these HCWs and status of return to work were captured by the infection control team in a systematic manner.

ELIGIBILITY:
Inclusion Criteria:

* All full time staff members of the private hospital

Exclusion Criteria:

* History of COVID-19 before 2022

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All full time staff members of the private hospital
Sampling Method: Probability Sample
Enrollment: 3167 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
COVID-19 Infection | During 1 February - 31 March 2022
  Number of participants with COVID-19 infected
Number of days return to work after COVID-19 infection | During 1 February - 31 March 2022
  Number of days return to work after COVID-19 infection

CONTACTS AND LOCATIONS:
Overall Officials: Jonpaul Sze Tsing Zee, MBChB, Principal Investigator — Hong Kong Sanatorium & Hospital
Locations (1):
- Hong Kong Sanatorium & Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No